CLINICAL TRIAL: NCT06183528
Title: Effects of Pericapsular Nerve Group Block on Postoperative Recovery for Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Ass prof, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UERH-AR-ZT-02
Record Dates: First submitted 2023-11-30; First posted 2023-12-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Analgesia; Postoperative Pain, Acute
Keywords: Multimodal analgesia; pericapsular nerve group block; total hip arthroplasty; spinal anesthesia
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: This prospective randomised controlled study included a total of 60 patients aged 40-85 years who underwent THA surgery under spinal anaesthesia. Patients were divided into two groups as PENG block and non-PENG block (control group).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Active Comparator): PENG block was placed in the fascial plane between the pseudotendon and pubic ramus with USG in-plane technique, 20 ml of 0.5% bupivacaine was administered after spinal anaesthesia.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block
- non-PENG group (Placebo Comparator): group non-PENG, surgery was started without PENG block after spinal anaesthesia.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — With ultrasonography-guided PENG block, the femoral, obturator and accessory obturator nerve branches that provide sensory innervation of the anterior surface of the hip joint capsule are blocked .

SUMMARY:
The hypothesis of this study is that patients who undergo PENG block in before Total Hip Artroplasthy (THA) surgery with spinal anesthesia will have reduced postoperative pain scores, less need for opioid analgesics and earlier mobilisation.

DETAILED DESCRIPTION:
This prospective randomised controlled study included a total of 60 patients aged 40-85 years who underwent THA surgery under spinal anaesthesia. Patients were divided into two groups as PENG block (n:30) and non-PENG block (n:30). PENG block was placed in the fascial plane between the pseudotendon and pubic ramus with USG in-plane technique, 20 ml of 0.5% bupivacaine was administered and surgery was initiated. The primary outcome of the study was to investigate the effect of preoperative PENG block application on postoperative pain, opioid requirement, mobilisation time, hip joint patency and length of hospital stay in patients undergoing THA surgery. The secondary outcome was to investigate the effect of PENG block on perioperative haemodynamics and postoperative side effects.

For multimodal analgesia, 10 ml 0.5% bupivacaine + 10 ml 2% lidocaine is infiltrated into the surgical wound incision line by the surgical team at the end of surgery. After tramadol 50 mg loading with PCA device, a basal rate of 5-10 mg/hour (20 mg bolus dose + 30 minutes lock time) is given with paracetamol 10 mg/kg iv (8 hours interval).

ELIGIBILITY:
Inclusion Criteria:

* THA performed by posterior approach
* 40-85 age range
* ASA 1-3

Exclusion Criteria:

Under 40 years of age, over 85 years of age,

* ASA 4 and above,
* Cognitive impairment (Alzheimer's disease, dementia, delirium etc.),
* Hip fracture,
* Application site infection,
* Allergy to local anaesthetic agents,
* Patients are non-consenting patients.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | recovery room 30 min, 12., 24. and 48. hours in the postoperative period
  VAS pain score
mobilisation time | 24 -48 hours
  walking 5 steps with walker
hip joint patency | 24. hours
  Measurement of joint movement angle with goniometer (angle)
total opioid consumption | 48 hours
  Tramadol total usage (mg)

SECONDARY OUTCOMES:
PENG block side effects | The first 48 hours after performing the PENG block
  motor block, nausea, vomiting, anaphylaxis, nerve damage
Perioperative haemodynamic data | T1: 30 minutes (min) after spinal anesthesia, T2: at the end of the surgical procedure, T3: at 30 minutes after recovery
  heart rate, mean arterial pressure
length of hospital stay | day
  hospitalization and discharge time for surgery

CONTACTS AND LOCATIONS:
Overall Officials: zeliha tuncel, Study Director — Ümraniye Training and Education hospital
Locations (1):
- UmraniyeERH, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No